CLINICAL TRIAL: NCT07099404
Title: Parathyroid Adenoma Detection With Rubidium Chloride Imaging: A Proof-of-Concept Study
Brief Title: Parathyroid Adenoma Detection With Rubidium-82 Imaging
Acronym: PARAGON
Status: Not yet recruiting | Type: Observational
Sponsor: Matthieu Pelletier-Galarneau, MD MSc (Other)
Responsible Party: Sponsor-Investigator, Matthieu Pelletier-Galarneau, MD MSc, Chief of the Nuclear Medicine Department, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Other Study IDs: MP-33-2025-3547
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Parathyroid Adenomas; Hyperparathyroidism, Primary
Keywords: Parathyroid adenomas, Rubidium-82
MeSH Terms: conditions — Parathyroid Neoplasms; Hyperparathyroidism, Primary | interventions — Rubidium-82

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PET/CT imaging with rubidium-82 — PET imaging of the neck will be started immediately before infusion of 10 Megabecquerels per kilograms of rubidum-82 over 30 seconds. The acquisition will last 10 minutes. This will be followed by a non-contrast low-dose CT of the neck for localization and attenuation correction.
  Other Names: Rubidium-82; PET/CT

SUMMARY:
Assess the uptake of rubidium-82 in parathyroid adenomas.

DETAILED DESCRIPTION:
Parathyroid adenomas demonstrate uptake of rubidium-82 chloride and can be detected with PET imaging.

The investigators aim to describe the uptake pattern of rubidium-82 chloride in parathyroid adenomas as well as compare the uptake pattern of rubidium-82 chloride to that of 18F-fluorocholine in patients with parathyroid adenoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18y
2. Ability to undergo imaging logistics
3. Ability to provide informed consent
4. Biochemical evidence of primary hyperparathyroidism
5. Documented parathyroid adenoma on prior 18F-fluorocholine imaging

Exclusion Criteria:

1. Normocalcemic primary hyperparathyroidism
2. Breastfeeding or pregnancy
3. Claustrophobia or inability to undergo imaging logistics
4. Any other history, condition, therapy, or uncontrolled intercurrent illness, which could in the opinion of the investigator affect compliance with study requirements or which would make the participant unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 participants with a diagnosis of primary parathyroid adenoma who have previously undergone 18F-fluorocholine imaging will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Uptake pattern of rubidium-82 in parathyroid adenomas | 3 months
  Rudibium-82 uptake will be assessed using Maximum Standardized Uptake Value (SUVmax) and target-to-background ratios (TBR). TBR is calculated by dividing a lesion SUVmax by the mean SUV (SUVmean) or the blood pool. Maximum Standardized Uptake Value (SUVmax) and target-to-background (TBR) will be presented as median with interquartile range as well as minimum and maximum values.

SECONDARY OUTCOMES:
Comparison between the uptakes of rubidium-82 and 18F-fluorocholine in patients with parathyroid adenomas | 3 months
  Radioactive tracer uptake will be compared between Rudibium-82 and 18F-Fluorocholine. Uptake will be assessed using Maximum Standardized Uptake Value (SUVmax) and target-to-background ratios (TBR). TBR is calculated by dividing a lesion SUVmax by the mean SUV (SUVmean) or the blood pool. Maximum Standardized Uptake Value (SUVmax) and target-to-background (TBR) will be presented as median with interquartile range as well as minimum and maximum values.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Montreal Heart Institute, Montreal, Quebec
  - Montreal Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No